CLINICAL TRIAL: NCT04056260
Title: Oncologic Safety of Sentinel Lymph Node-guided Lymph Node Dissection Using ICG-NIR Laparoscopy in Gastric Cancer
Brief Title: ICG-NIR Guided Lymph Node Dissection in Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ho Seok Seo (Other)
Responsible Party: Sponsor-Investigator, Ho Seok Seo, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDR-01
Record Dates: First submitted 2019-08-11; First posted 2019-08-14 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Stomach Neoplasm
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICG injection (Experimental): ICG 0.5mg/ml x 0.5ml x 4 sites
  Interventions: Procedure: ICG-NIR guided surgery

INTERVENTIONS:
Procedure: ICG-NIR guided surgery — ICG 0.5mg/ml x 0.5ml x 4 sites injection through intra-operative endoscopy

SUMMARY:
As the survival rate of patients with gastric cancer has increased, there has been a growing interest in interventions that improve postoperative quality of life. Therefore minimally invasive surgery or endoscopic resection has been performed much more frequently. However, adequate lymph node dissection is important as well. The aim of the study is to identify the feasibility of indocyanine green - near infra-red (ICG-NIR) guided sentinel lymph node dissection for the treatment of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* dignosed gastric adenocarcinoma
* tumor: size 4cm or smaller
* depth of invasion: mucosa, submucosa, proper muscle
* candidates of laparoscopic radical gastrectomy
* informed consent

Exclusion Criteria:

* metachronous malignancy
* number of tumors: 2 or more
* remnant gastric cancer
* indication for endoscopic resection
* history of chemotherapy or radiation therapy
* pregnancy
* allergy to ICG
* metastatic gastric cancer

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Estimated)
Dates: Start 2020-03-20 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity | 1 month
  sensitivity and specificity of ICG-NIR guided lymph node dissection